CLINICAL TRIAL: NCT04763161
Title: Immuno-inflammation in the Acute Phase of an Ischaemic Cerebral Accident Managed by Decompressive Hemicraniectomy: a Case-control Study
Acronym: NEUTROSURGERY
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: BMR_2021_2
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Patients suffering from malignant sylvian ischaemic cerebral accident and treated with decompressive hemicraniectomy.
  Intervention is decompressive hemicraniectomy in the context of a malignant sylvian ischaemic cerebral
  Interventions: Procedure: Decompressive hemicraniectomy
- Control group: Patients not suffering from AIC, hospitalised in neurosurgery for another reason,
  Patients to be opered on which cranial, meningeal, vascular (branch of the middle meningeal artery) or cerebral bone tissue is not preserved during the surgical approach.
  Interventions: Procedure: neurosurgical operation

INTERVENTIONS:
Procedure: Decompressive hemicraniectomy — Decompressive hemicraniectomy in the context of a malignat sylvian ischaemic cerebral accident
  Groups: Experimental group
Procedure: neurosurgical operation — neurosurgical operation on which cranial, meningeal, vascular (branch of the middle meningeal artery) or cerebral bone tissue is not preserved during the surgical approach.
  Groups: Control group

SUMMARY:
The objective of the NEUTROSURGERY study is to describe the local and locoregional immuno-inflammatory activity in patients suffering from malignant sylvian ischaemic cerebral accident and treated with decompressive hemicraniectomy compared to a control population of patients to be operated on in neurosurgery for another neurosurgical pathology.

ELIGIBILITY:
Inclusion Criteria Patients:

* Collegial indication given by a neurologist, a neuroreanimator and a neurosurgeon for HD in the context of a malignant sylvian AIC.

Inclusion Criteria Control:

- For neurosurgical operations in which cranial, meningeal, vascular (branch of the middle meningeal artery) or cerebral bone tissue is not preserved during the surgical approach.

Non-inclusion Criteria Patients:

* HD carried out in a context of acute cerebral haemorrhage
* Pre-existing neurological disability: modified Rankin score > 2
* Patient benefiting from a legal protection measure

Non-inclusion Criteria Controls:

* Patient to be operated on for an acute vascular condition: meningeal haemorrhage, subdural or extradural haemorrhage, intra parenchymal haemorrhage.
* Patient operated on for an osteomeningeal pathology present at the approach site.
* Patient operated on for an infectious cranial or neuro-meningeal pathology.
* Patient to be operated on as a result of an intracranial traumatic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population concerns patients suffering from malignant sylvian ischaemic cerebral accident and treated with decompressive hemicraniectomy. Eligibility will be assessed as soon as the first results of the MRI or brain scan carried out as part of the thrombolysis alert by the interventional neurologist or neuroradiologist triggering the treatment, in front of a large ischaemic cerebral accident (>145 ml).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-08-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
neutrophil polynuclear cells levels | Day 0